CLINICAL TRIAL: NCT04439006
Title: Randomized Double-Blind Phase 2 Trial of Ibrutinib Versus Standard Treatment for COVID-19 Illness Requiring Hospitalization With Safety Lead-In
Brief Title: Ibrutinib for the Treatment of COVID-19 in Patients Requiring Hospitalization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer Woyach (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Woyach, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20135; NCI-2020-03341 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Aplastic Anemia; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Monoclonal B-Cell Lymphocytosis; Monoclonal Gammopathy of Undetermined Significance; Myelodysplastic Syndrome; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — Anemia, Aplastic; Hematologic Neoplasms; Monoclonal Gammopathy of Undetermined Significance; Myelodysplastic Syndromes | interventions — Practice Guidelines as Topic; Standard of Care; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-7. Treatment repeats every 7 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients who remain hospitalized or are re-admitted after 2 cycles may receive an additional 2 cycles per physician's discretion.
  Interventions: Drug: Ibrutinib
- Arm B (usual care) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm B (usual care)
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
  Arms: Arm A (ibrutinib)

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of ibrutinib and how well it works in treating patients with COVID-19 requiring hospitalization. Ibrutinib may help improve COVID-19 symptoms by lessening the inflammatory response in the lungs, while preserving overall immune function. This may reduce the need to be on a ventilator to help with breathing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and tolerability of administering ibrutinib in COVID-19 infected patients and determining the recommended phase 2 dose (RP2D). (Phase Ib) II. To determine whether ibrutinib administration (Arm A) in cancer patients can diminish the need for artificial ventilation (mechanical ventilation, bilevel positive airway pressure [BiPAP] or extracorporeal membrane oxygenation [ECMO]) or death due to COVID-19 as compared to untreated control population receiving standard therapy (antiviral, chloroquine, hydroxychloroquine, cytokine blocking peptides or small molecules) (Arm B). (Phase II)

SECONDARY OBJECTIVES:

I. To determine the time to defervescence (oral temperature < 100.5 degrees Fahrenheit [F] for a 48 hour time period) among patients treated with ibrutinib (Arm A) versus control population receiving standard (Arm B) therapy.

II. To determine time to clinical resolution of need for supplemental oxygen (i.e. maintenance of oxygen saturation of 93% or greater on room air with ambulation).

III. To determine rate of intensive care unit (ICU) admission and length of ICU admission for patients treated with ibrutinib (Arm A) versus control population receiving standard therapy (Arm B).

IV. To determine rate of shock requiring vasopressor support for patients treated with ibrutinib (Arm A) versus control population receiving standard therapy (Arm B).

V. To determine the rate of secondary infection (bacterial, fungal, viral) for patients treated with ibrutinib (Arm A) versus control population receiving standard therapy (Arm B).

VI. To determine the time to hospital discharge for patients treated with ibrutinib (Arm A) versus control population receiving standard therapy (Arm B).

VII. To determine time to hospital discharge and rate of death for patients who cross over to ibrutinib (Arm A) from standard therapy (Arm B).

VIII. To determine grade 3 or higher toxicity observed in patients treated with ibrutinib (Arm A) versus control population receiving standard therapy (Arm B).

IX. To determine time to mechanical ventilation, the number of days of mechanical ventilation per patient and total observed in patients treated with ibrutinib (Arm A) versus control population receiving standard therapy (Arm B).

EXPLORATORY OBJECTIVES:

I. To examine the impact of baseline clinical features (e.g. type of cancer, active therapy), duration of symptoms prior to admission and laboratory features (e.g. T cell count) on outcome for patients treated on this therapeutic study.

II. To determine the proportion of patients with viral clearance at end of ibrutinib therapy, time of hospital discharge and follow up thereafter among patients treated with ibrutinib (Arm A) versus control (Arm B) treatment.

III. To determine the time and proportion of patients who develop immunoglobulin (Ig)M and IgG levels toward SARS-coronavirus (CoV)-2 treated with ibrutinib (Arm A) versus control treatment (Arm B).

IV. To examine immune cell subsets for absolute number, activation, exhaustion markers, and presence of maturation arrest (natural killer [NK] cells) at baseline and over time among patients treated with ibrutinib (Arm A) versus control (Arm B) treatment.

V. To examine T-cell repertoire over time among patients treated with ibrutinib (Arm A) versus control (Arm B) treatment.

VI. To determine the influence of epigenetic age, clonal hematopoiesis, and monoclonal B cell lymphocytosis (MBL) on treatment outcome.

VII. To determine serial change in inflammatory markers as CRP, ferritin, D-dimer and cytokines including IL6, IL1B, and TNF-alpha serum levels over time among patients treated with ibrutinib (Arm A) versus control (Arm B) treatment.

OUTLINE: This is a phase Ib, dose-escalation study followed by a phase II study.

The first 12 patients will all receive ibrutinib. In the randomized part, patients are randomized to 1 of 2 arms.

ARM A: Patients receive ibrutinib orally (PO) once daily (QD) on days 1-7. Treatment repeats every 7 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients who remain hospitalized or are re-admitted after 2 cycles may receive an additional 2 cycles per physician's discretion.

ARM B: Patients receive usual care. Patients who meet the requirement of mechanical ventilation may cross-over to Arm A.

After completion of study treatment, patients are followed up for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* History or active diagnosis of cancer (solid or hematologic) or precursor of cancer (monoclonal gammopathy of undetermined significance [MGUS]), monoclonal B lymphocytosis (MBL), aplastic anemia or myelodysplastic syndrome) that is associated with immune suppression
* Hospitalization for confirmed polymerase chain reaction (PCR) positive COVID-19 infection
* Patients with evidence of pulmonary involvement who meet any of the followings; presence of infiltrates on chest X-ray or computed tomography (CT) scan or need for supplemental oxygen < 8 L nasal cannula or pulse oximetry < 94% on room air
* Creatinine clearance >= 25 ml/min by Cockcroft-Gault equation
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Absolute neutrophil count (ANC) >= 1000/mm^3 independent of growth factor support
* Platelets >= 50,000/mm^3
* Ability to swallow capsules
* Ability to provide informed consent indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study

Exclusion Criteria:

* New-onset malignancy requiring urgent initiation of systemic chemotherapy
* Active uncontrolled systemic bacterial or fungal or other viral infection
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon)
* Currently receiving BTK inhibitor therapy
* Actively receiving anti-cancer therapy (other than hormonal therapies). All anti-cancer therapy (except hormonal therapies) must be stopped at the time of screening; can be resumed as soon as ibrutinib is discontinued. Significantly T cell suppressive chemotherapy (defined as requiring PJP prophylaxis per standard guidelines) is not allowed for 3 months prior to enrollment.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional classification requirement for mechanical ventilation at screening
* Known bleeding disorders (e.g., Von Willebrand's disease, platelet storage pool disorders, or hemophilia)
* Stroke or intracranial hemorrhage within 6 months of screening
* Major surgery or non-healing wound within 4 weeks of enrollment
* Concomitant administration of prohibited medications
* Known history of human immunodeficiency virus (HIV), or active hepatitis B or C infection
* Disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption (malabsorption syndrome, resection of the small bowel, poorly controlled inflammatory bowel disease, etc.)
* Requires chronic treatment with strong CYP3A inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with diminished respiratory failure and death | During hospitalization for COVID-19 infection or within 30 days of registration
  Associations between baseline characteristics and the primary endpoint will be evaluated with logistic regression, adjusting for arm. These analyses will be largely descriptive, as a result of a limited sample size.
Death | During hospitalization for COVID-19 infection or within 30 days of registration

SECONDARY OUTCOMES:
Time from study initiation to 48 hours fever-free | Up to 14 days
  Fever-free will be assessed by a temperature of < 100.5 degrees Fahrenheit orally. Will be estimated for each arm using the method of Kaplan-Meier. Medians estimates and/or estimates at specific time points will be provided with 95% confidence intervals.
Duration of hospitalization | Up to 14 days
  Will be estimated for each arm using the method of Kaplan-Meier. Medians estimates and/or estimates at specific time points will be provided with 95% confidence intervals.
Time in intensive care unit (ICU) | Up to 14 days
Time to ICU admission | Up to 14 days
Number of days requiring supplemental oxygen | Up to 14 days
Total days of mechanical ventilation | Up to 14 days
Time to mechanical ventilation | Up to 14 days
Shock and need for pressure support | Up to 14 days
Incidence of any infection (viral, fungal, bacterial) | Up to 14 days
Time to clinical resolution | Up to 14 days
Incidence of grade 3 or higher adverse events | Up to 12 months
  Adverse events will be summarized by grade, type, and attribution (regardless of attribution and treatment-related) for each arm.
At the end of therapy (day 14) | Up to 14 days
  The proportion of patients with viral clearance at the time of hospital discharge will be estimated with 95% confidence intervals for each arm.
Time to viral clearance | Up to 12 months
  Will be estimated for each arm using the method of Kaplan-Meier. Medians estimates and/or estimates at specific time points will be provided with 95% confidence intervals.
Survival | Up to12 months
  Patients will be followed for up to 12 months or until death or withdrawal of study consent for further follow-up. Following hospitalization, study visits will be telephone or video encounters.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Woyach, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04439006/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT04439006/ICF_000.pdf